CLINICAL TRIAL: NCT02983552
Title: Binocular Dig Rush Game Treatment for Amblyopia
Acronym: ATS20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS20; 2U10EY011751 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-12-06 (Estimated); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Amblyopia
Keywords: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binocular Computer Game Treatment (Experimental): Binocular computer game treatment is defined as playing a Dig Rush application on an iPad® 1 hour per day, 5 days per week for 8 weeks in addition to continued spectacle correction (if required)
  Interventions: Other: iPad®
- Continued Spectacle Correction (Active Comparator): Continued spectacle correction is defined as wearing appropriate spectacle correction (if required) for all waking hours, 7 days per week for 8 weeks.
  Interventions: Other: Spectacle correction

INTERVENTIONS:
Other: iPad® — Binocular therapy using a Dig Rush application on an iPad®
  Arms: Binocular Computer Game Treatment
Other: Spectacle correction — Spectacle correction for all waking hours, 7 days per week
  Arms: Continued Spectacle Correction

SUMMARY:
To compare the efficacy of 1 hour/day of binocular game play 5 days per week plus spectacle correction with spectacle correction only, for treatment of amblyopia in children 4 to <13 years of age.

DETAILED DESCRIPTION:
The purpose of the study is to compare the efficacy of 1 hour/day of binocular game play 5 days per week plus spectacle correction with spectacle correction only, for treatment of amblyopia in children 4 to <13 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 to <13 years
2. Amblyopia associated with strabismus, anisometropia, or both (previously treated or untreated)

   1. Criteria for strabismic amblyopia: At least one of the following must be met:

      * Presence of a heterotropia on examination at distance or near fixation (with or without optical correction, must be no more than 5pd by SPCT at near fixation (see #6 below)
      * Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia)
   2. Criteria for anisometropia: At least one of the following criteria must be met:

      * ≥1.00 D difference between eyes in spherical equivalent
      * ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes
   3. Criteria for combined-mechanism amblyopia: Both of the following criteria must be met:

      * Criteria for strabismus are met (see above)
      * ≥1.00 D difference between eyes in spherical equivalent OR ≥1.50 D difference in astigmatism between corresponding meridians in the two eyes
3. No amblyopia treatment other than optical correction in the past 2 weeks (patching, atropine, Bangerter, vision therapy, binocular treatment)
4. Requirements for required refractive error correction (based on a cycloplegic refraction completed within the last 7 months):

   * Hypermetropia of 2.50 D or more by spherical equivalent (SE)
   * Myopia of amblyopic eye of 0.50D or more SE
   * Astigmatism of 1.00D or more
   * Anisometropia of more than 0.50D SE

   NOTE: Subjects with cycloplegic refractive errors that do not fall within the requirements above for spectacle correction may be given spectacles at investigator discretion but must follow the study-specified prescribing guidelines, as detailed below.
   1. Spectacle prescribing instructions referenced to the cycloplegic refraction completed within the last 7 months:

      * SE must be within 0.50D of fully correcting the anisometropia.
      * SE must not be under corrected by more than 1.50D SE, and reduction in plus sphere must be symmetric in the two eyes.
      * Cylinder power in both eyes must be within 0.50D of fully correcting the astigmatism.
      * Axis must be within +/- 10 degrees if cylinder power is ≤1.00D, and within +/- 5 degrees if cylinder power is >1.00D.
      * Myopia must not be undercorrected by more than 0.25D or over corrected by more than 0.50D SE, and any change must be symmetrical in the two eyes.
   2. Spectacle correction meeting the above criteria must be worn:

      * For at least 16 weeks OR until VA stability is documented (defined as <0.1 logMAR change by the same testing method measured on 2 consecutive exams at least 8 weeks apart).
      * For determining VA stability (non-improvement):

        * The first of two measurements may be made 1) in current spectacles, or 2) in trial frames with or without cycloplegia or 3) without correction (if new correction is prescribed),
        * The second measurement must be made without cycloplegia in the correct spectacles that have been worn for at least 8 weeks.
        * Note: since this determination is a pre-study procedure, the method of measuring VA is not mandated.
5. VA, measured in each eye without cycloplegia in current spectacle correction (if applicable) within 7 days prior to randomization using the ATS-HOTV VA protocol for children < 7 years and the E-ETDRS VA protocol for children ≥ 7 years on a study-approved device displaying single surrounded optotypes, as follows:

   1. VA in the amblyopic eye 20/40 to 20/200 inclusive (ATS-HOTV) or 33 to 72 letters (E-ETDRS)
   2. VA in the fellow eye 20/25 or better (ATS-HOTV) or ≥ 78 letters (E-ETDRS)
   3. Interocular difference ≥ 3 logMAR lines (ATS-HOTV) or ≥ 15 letters (E-ETDRS)
6. Heterotropia with a near deviation of ≤ 5∆ (measured by SPCT) in habitual correction (Angles of ocular deviation >5∆ are not allowed because large magnitudes of the deviation would compromise successful playing of the game.)
7. Subject is able to play the Dig Rush game (at least level 3) on the study iPad under binocular conditions (with red-green glasses). Subject must be able to see both the red "diggers" and blue "gold carts" when contrast for the non-amblyopic eye is at 20%.
8. Investigator is willing to prescribe computer game play, or continued spectacle wear per protocol.
9. Parent understands the protocol and is willing to accept randomization.
10. Parent has phone (or access to phone) and is willing to be contacted by Jaeb Center staff or other study staff.
11. Relocation outside of area of an active PEDIG site for this study within the next 8 weeks is not anticipated.

Exclusion Criteria:

1. Prism in the spectacle correction at time of enrollment (eligible only if prism is discontinued 2 weeks prior to enrollment).
2. Myopia greater than -6.00D spherical equivalent in either eye.
3. Previous intraocular or refractive surgery.
4. Any treatment for amblyopia (patching, atropine, Bangerter filter, vision therapy or previous binocular treatment) during the past 2 weeks. Previous amblyopia therapy is allowed regardless of type, but must be discontinued at least 2 weeks prior to enrollment.
5. Ocular co-morbidity that may reduce VA determined by an ocular examination performed within the past 7 months (Note: nystagmus per se does not exclude the subject if the above VA criteria are met).
6. No Down syndrome or cerebral palsy
7. No severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Subjects with mild speech delay or reading and/or learning disabilities are not excluded.
8. Subject has demonstrated previous low compliance with binocular treatment and/or spectacle treatment (as assessed informally by the investigator)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Manny, OD, PhD, Study Chair — University of Houston College of Optometry; Jonathan Holmes, MD, Study Chair — Mayo Clinic
Locations (62):
- United States (61):
  - UAB Pediatric Eye Care; Birmingham Health Care, Birmingham, Alabama
  - Midwestern University Eye Institute, Glendale, Arizona
  - University Eye Center at Ketchum Health, Anaheim, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Saddleback Eye Medical Associates, Mission Viejo, California
  - Western University College of Optometry, Pomona, California
  - Yale University, New Haven, Connecticut
  - Nova Southeastern University College of Optometry, The Eye Institute, Fort Lauderdale, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - The Emory Eye Center, Atlanta, Georgia
  - St Luke's Hospital, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - Ticho Eye Associates, Chicago Ridge, Illinois
  - Progressive Eye Care, Lisle, Illinois
  - Advanced Vision Center, Schaumburg, Illinois
  - Pediatric Eye Associates, Wilmette, Illinois
  - Indiana School of Optometry, Bloomington, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Wilmer Eye Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Michigan College of Optometry at Ferris State Univ, Big Rapids, Michigan
  - Helen DeVos Children's Hospital Pediatric Ophthalmology, Grand Rapids, Michigan
  - Pediatric Ophthalmology, P.C., Grand Rapids, Michigan
  - University of Minnesota-Minnesota Lions Children's Eye Clinic, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Saint Louis University Institute, St Louis, Missouri
  - St. Louis Children's Hospital Eye Center, St Louis, Missouri
  - U of MO St. Louis College of Optometry, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Concord Ophthalmologic Associates, Concord, New Hampshire
  - Michael F. Gallaway, O.D., P.C., Marlton, New Jersey
  - State University of New York, College of Optometry, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Eye Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Pediatric Ophthalmology Associates, Inc., Columbus, Ohio
  - The Ohio State University College of Optometry, Columbus, Ohio
  - Eye Care Associates, Inc., Poland, Ohio
  - Dean A. McGee Eye Institute, University of Oklahoma, Oklahoma City, Oklahoma
  - Pacific University College of Optometry, Portland, Oregon
  - OHSU Casey Eye Institute, Portland, Oregon
  - Pediatric Ophthalmology of Erie, Erie, Pennsylvania
  - Conestoga Eye, Lancaster, Pennsylvania
  - Pediatric Eye Specialists, Chattanooga, Tennessee
  - Southern College of Optometry, Memphis, Tennessee
  - Texas Children's Hospital - Dept. Of Ophthalmology, Houston, Texas
  - University of Houston College of Optometry, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Houston Eye Associates, The Woodlands, Texas
  - Virginia Pediatric Eye Center, Norfolk, Virginia
  - Seattle Children's Hospital, University of Washington, Seattle, Washington
  - Northwest Pediatric Ophthalmology, P.S., Spokane, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
  - Marshall University, Huntington, West Virginia
  - University of Wisconsin, University Station, Madison, Wisconsin
  - Snowy Range Vision Center, Laramie, Wyoming
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group; Holmes JM, Manny RE, Lazar EL, Birch EE, Kelly KR, Summers AI, Martinson SR, Raghuram A, Colburn JD, Law C, Marsh JD, Bitner DP, Kraker RT, Wallace DK. A Randomized Trial of Binocular Dig Rush Game Treatment for Amblyopia in Children Aged 7 to 12 Years. Ophthalmology. 2019 Mar;126(3):456-466. doi: 10.1016/j.ophtha.2018.10.032. Epub 2018 Oct 22. PMID 30352226
- [Derived] Manny RE, Holmes JM, Kraker RT, Li Z, Waters AL, Kelly KR, Kong L, Crouch ER, Lorenzana IJ, Alkharashi MS, Galvin JA, Rice ML, Melia BM, Cotter SA; Pediatric Eye Disease Investigator Group. A Randomized Trial of Binocular Dig Rush Game Treatment for Amblyopia in Children Aged 4 to 6 Years. Optom Vis Sci. 2022 Mar 1;99(3):213-227. doi: 10.1097/OPX.0000000000001867. PMID 35086119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 138 is the number of subjects from the older cohort study. 182 is the number of subjects from the younger cohort.
Groups:
- Binocular Computer Game Treatment- Older Cohort; Binocular Computer Game Treatment- Younger Cohort: Binocular computer game treatment is defined as playing a Dig Rush application on an iPad® 1 hour per day, 5 days per week for 8 weeks in addition to continued spectacle correction (if required)
  iPad®: Binocular therapy using a Dig Rush application on an iPad®
- Continued Spectacle Correction- Older Cohort; Continued Spectacle Correction- Younger Cohort: Continued spectacle correction is defined as wearing appropriate spectacle correction (if required) for all waking hours, 7 days per week for 8 weeks.
  Spectacle correction: Spectacle correction for all waking hours, 7 days per week
Period: Overall Study
Arm/Group | Binocular Computer Game Treatment- Older Cohort | Continued Spectacle Correction- Older Cohort | Binocular Computer Game Treatment- Younger Cohort | Continued Spectacle Correction- Younger Cohort
Started | 69 | 69 | 92 | 90
4 Week Visit | 69 | 67 | 85 | 84
8 Week Visit | 67 | 68 | 85 | 84
16 Week Visit (The 16 week visit was elective for those who were originally assigned to continued spectacle correction. After completing 8 weeks of continued spectacle correction, participants were able to complete 8 weeks of binocular therapy. Values are not provided for the binocular computer game treatment cohorts as this visit was not applicable.) | 0 (The 16 week visit was elective for those who were originally assigned to continued spectacle correction. After completing 8 weeks of continued spectacle correction, participants were able to complete 8 weeks of binocular therapy. Values are not provided for the binocular computer game treatment cohorts as this visit was not applicable.) | 66 | 0 (The 16 week visit was elective for those who were originally assigned to continued spectacle correction. After completing 8 weeks of continued spectacle correction, participants were able to complete 8 weeks of binocular therapy. Values are not provided for the binocular computer game treatment cohorts as this visit was not applicable.) | 72
Completed | 69 | 67 | 92 | 90
Not Completed | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Binocular Computer Game Treatment Older Cohort; Binocular Computer Game Treatment Younger Cohort: Binocular computer game treatment is defined as playing a Dig Rush application on an iPad® 1 hour per day, 5 days per week for 8 weeks in addition to continued spectacle correction (if required)
  iPad®: Binocular therapy using a Dig Rush application on an iPad®
- Continued Spectacle Correction Older Cohort; Continued Spectacle Correction Younger Cohort: Continued spectacle correction is defined as wearing appropriate spectacle correction (if required) for all waking hours, 7 days per week for 8 weeks.
  Spectacle correction: Spectacle correction for all waking hours, 7 days per week
- Total: Total of all reporting groups
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort | Total
Number analyzed (Participants) | 69 | 69 | 92 | 90 | 320
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 69 | 69 | 92 | 90 | 320
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (1.6) | 9.6 (1.5) | 5.8 (0.7) | 5.7 (0.7) | 7.4 (2.2)
Age, Customized [Count of Participants; unit: Participants]
  Age Range: 7 to <10 years | 45 | 45 | 0 | 0 | 90
  Age Range: 10 to <13 years | 24 | 24 | 0 | 0 | 48
  Age Range: 4 to <5 years | 0 | 0 | 12 | 17 | 29
  Age Range: 5 to <6 years | 0 | 0 | 39 | 41 | 80
  Age Range: 6 to <7 years | 0 | 0 | 41 | 32 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 50 | 46 | 161
  Male | 39 | 34 | 42 | 44 | 159
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 55 | 75 | 74 | 254
  Black/African American | 3 | 2 | 2 | 5 | 12
  Hispanic | 9 | 8 | 12 | 8 | 37
  Asian | 6 | 1 | 1 | 2 | 10
  More than one race | 1 | 2 | 2 | 1 | 6
  Unknown/not reported | 0 | 1 | 0 | 0 | 1
Prior Amblyopia Treatment [Count of Participants; unit: Participants]
  None | 4 | 2 | 33 | 32 | 71
  Patching | 34 | 36 | 39 | 40 | 149
  Atropine | 0 | 1 | 2 | 2 | 5
  Patching/Atropine | 26 | 21 | 15 | 15 | 77
  Patching/Other | 3 | 2 | 1 | 1 | 7
  Patching/Atropine/Other | 2 | 7 | 2 | 0 | 11
Prior Binocular Treatment [Count of Participants; unit: Participants] | 1 | 4 | 0 | 0 | 5
Distance Amblyopic-eye VA (Letter Score) [Count of Participants; unit: Participants]
  20/160 | 2 | 2 | 2 | 3 | 9
  20/125 | 3 | 3 | 7 | 3 | 16
  20/100 | 8 | 8 | 3 | 4 | 23
  20/80 | 10 | 17 | 9 | 9 | 45
  20/63 | 19 | 14 | 24 | 24 | 81
  20/50 | 11 | 10 | 27 | 26 | 74
  20/40 | 16 | 15 | 19 | 19 | 69
  20/200 | 0 | 0 | 1 | 2 | 3
Distance Amblyopic-eye VA [Mean (Standard Deviation); unit: logMAR] | 0.50 (0.16) | 0.52 (0.16) | 0.48 (0.16) | 0.48 (0.17) | 0.49 (0.16)
Distance Fellow-eye VA [Mean (Standard Deviation); unit: logMAR] | -0.058 (0.079) | -0.058 (0.074) | 0.002 (0.083) | -0.003 (0.085) | -0.025 (0.086)
Interocular Difference (Lines) [Mean (Standard Deviation); unit: Lines] | 5.57 (1.83) | 5.75 (1.86) | 4.80 (4.86) | 1.71 (1.70) | 5.19 (1.81)
Stereoacuity: Nil [Count of Participants; unit: Participants] | 33 | 33 | 29 | 28 | 123
Stereoacuity (Seconds of Arc) [Median (Full Range); unit: Seconds of Arc] — Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (measured as seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool (scores: 800, 400, 200, 100, 60 and 40) stereoacuity test methods as previously described. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores (Nil was assigned a score of 4000) to the log scale to calculate descriptive statistics (reported as seconds of arc).
  Seconds of Arc | 2000 [40 to 4000] | 2000 [40 to 4000] | 800 [40 to 4000] | 800 [40 to 4000] | 2000 [40 to 4000]
Amblyopia Cause [Count of Participants; unit: Participants]
  Strabismus | 15 | 11 | 15 | 15 | 56
  Anisometropia | 27 | 39 | 61 | 54 | 181
  Combined-mechanism | 27 | 19 | 16 | 21 | 83
Distance SPCT: Maximum angle of deviation [Count of Participants; unit: Participants]
  Orthotropic | 47 | 50 | 73 | 76 | 246
  1 to 4 prism diopters | 18 | 15 | 15 | 11 | 59
  5 to 9 prism diopters | 2 | 2 | 3 | 2 | 9
  >=10 prism diopters | 2 | 2 | 1 | 1 | 6
Near SPCT: Maximum angle of deviation [Count of Participants; unit: Participants]
  Orthotropic | 44 | 47 | 72 | 75 | 238
  1 to 4 prism diopters | 25 | 22 | 20 | 15 | 82
Amblyopic-eye Spherical Equivalent (Diopters) [Mean (Standard Deviation); unit: Diopters] | 4.35 (2.42) | 4.40 (2.28) | 4.49 (1.75) | 4.45 (2.76) | 4.43 (2.32)
Fellow-eye Spherical Equivalent (Diopters) [Mean (Standard Deviation); unit: Diopters] | 2.10 (2.12) | 2.22 (1.99) | 2.41 (1.67) | 2.67 (1.99) | 2.38 (1.93)
Spherical Equivalent Anisometropia (Diopters) [Mean (Standard Deviation); unit: Diopters] | 2.29 (1.79) | 2.27 (1.62) | 2.12 (1.52) | 2.25 (1.51) | 2.22 (1.59)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Amblyopic-eye Visual Acuity (VA) Older Cohort
Description: The primary objective is to compare the efficacy of 4 weeks of treatment with 1 hour/day of binocular game play 5 days per week plus spectacle correction to treatment with spectacle correction alone (control). Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the analyses in the older cohort, the level of VA is measured as letter scores (approximate range: 0 to 97 letters, lower scores indicate poorer VA) and change in VA from baseline is measured in letters (positive values indicate improvement), defined as the difference in letter scores between enrollment and follow-up.
  Adjusted values have been adjusted for amblyopic-eye visual acuity at randomization.
Time Frame: Baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: Letter score
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort
Number analyzed (Participants) | 69 | 67
Letter score
  Adjusted | 1.3 [0.1 to 2.6] | 1.7 [0.4 to 3.0]
  Unadjusted | 1.3 [0.1 to 2.6] | 1.7 [0.4 to 3.0]
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; A modified intent-to-treat analysis was performed using an ANCOVA model to compare the effectiveness of two treatments (2-sided hypothesis test), adjusting for baseline visual acuity. The primary outcome measure was change in amblyopic-eye VA from baseline to 4 weeks. A 2-sided 95% confidence interval (CI) was computed on the adjusted treatment group difference at 4 weeks. There was no imputation for missing data; Test type: Superiority; p = 0.71, ANOVA — a priori threshold for statistical significance: 2-sided type I error rate of 5%; Adjusted for baseline amblyopic-eye visual acuity; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.2 to 1.7] — A 2-sided 95% confidence interval was computed on the adjusted treatment group difference evaluating change in amblyopic-eye visual acuity from baseline to the 4 week visit

2. Primary Outcome: Mean Visual Acuity (VA) in Amblyopic-eye (Older Cohort)
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the analyses in the older cohort, the level of VA is measured as letter scores (approximate range: 0 to 97 letters, lower scores indicate poorer VA) and change in VA from baseline is measured in letters (positive values indicate improvement), defined as the difference in letter scores between enrollment and follow-up.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Letter score
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort
Number analyzed (Participants) | 69 | 67
Letter score | 26.6 (10.5) | 28.0 (10.7)

3. Primary Outcome: Mean Change in Amblyopic-eye Visual Acuity (VA) in Older Cohort
Description: as for outcome 2
Time Frame: Baseline and 8 weeks
Population: Two participants (1 per group) were not included with the 8-week visual acuity data. One participant in the control treatment group had visual acuity tested using a non-protocol method and another participant in the binocular treatment group completed the 8-week exam outside of the analysis window (49 to <105 days from randomization).
Measure: Mean (Full Range); unit: Letters
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort
Number analyzed (Participants) | 67 | 67
Letters
  Adjusted | 2.3 [0.7 to 3.9] | 2.4 [0.8 to 4.0]
  Unadjusted | 2.3 [0.6 to 4.0] | 2.4 [0.9 to 4.0]
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Test type: Superiority; Mean Difference (Final Values) = -0.1, 98.3% CI 2-sided [-2.4 to 2.1] — A 2-sided 98.3% confidence interval was computed on the adjusted treatment group difference evaluating change in amblyopic-eye visual acuity from baseline to the 8-week visit

4. Primary Outcome: Mean Visual Acuity (VA) in Amblyopic-eye (Older Cohort)
Description: as for outcome 2
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Letter score
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort
Number analyzed (Participants) | 67 | 67
Letter score | 25.9 (9.9) | 27.7 (10.4)

5. Primary Outcome: Mean Change in Amblyopic-eye Visual Acuity (VA) Younger Cohort
Description: The primary objective is to compare the efficacy of 4 weeks of treatment with 1 hour/day of binocular game play 5 days per week plus spectacle correction to treatment with spectacle correction alone (control). Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the analyses in the younger cohort, the level of VA is measured in logMAR (approximate range: -0.2 to 1.2, lower scores indicate better VA) and change in VA from baseline is measured in logMAR lines (positive values indicate improvement), defined as 10 times the difference in logMAR between enrollment and follow-up.
  Adjusted values have been adjusted for amblyopic-eye visual acuity at randomization.
Time Frame: baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: logMAR Lines
Arm/Group | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 85 | 84
logMAR Lines
  Adjusted | 1.0724 [0.8 to 1.4] | 0.6053 [0.3 to 0.9]
  Unadjusted | 1.0706 [0.8 to 1.4] | 0.6071 [0.3 to 0.9]

6. Primary Outcome: Mean Visual Acuity (VA) in Amblyopic-eye (Younger Cohort)
Description: Monocular distance visual acuity (VA) in current refractive correction (if required) in each eye by a certified examiner using the Electronic Early Treatment Diabetic Retinoscopy Study (E-ETDRS) visual acuity protocol for children ≥ 7 years on a study-certified acuity tester displaying single surrounded optotypes.
  For the analyses in the younger cohort, the level of VA is measured in logMAR (approximate range: -0.2 to 1.2, lower scores indicate better VA) and change in VA from baseline is measured in logMAR lines (positive values indicate improvement), defined as 10 times the difference in logMAR between enrollment and follow-up.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 85 | 84
LogMAR | 0.38 (0.22) | 0.42 (0.21)

7. Primary Outcome: Mean Change in Amblyopic-eye Visual Acuity (VA) in Younger Cohort
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: logMAR Lines
Arm/Group | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 85 | 84
logMAR Lines
  Adjusted | 1.2614 [1.0 to 1.6] | 0.9855 [0.7 to 1.3]
  Unadjusted | 1.2588 [1.0 to 1.6] | 0.9981 [0.7 to 1.3]

8. Primary Outcome: Mean Visual Acuity (VA) in Amblyopic-eye (Younger Cohort)
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 85 | 84
LogMAR | 0.36 (0.22) | 0.38 (0.22)

9. Secondary Outcome: VA Improvement at 4 Weeks Defined as a Binary Outcome
Description: A secondary analysis will estimate the proportion of subjects with amblyopic-eye VA improvement of ≥ 2 logMAR lines (≥ 10 letters if E-ETDRS) at 4 weeks after baseline.
Time Frame: At 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 85 | 84
Participants | 2 | 3 | 31 | 16
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Binomial regression was used for the treatment group comparison of the proportion of participants classified as improving 2 or more logMAR lines (10 or more letters if E-ETDRS) from baseline at the 4-week visit, adjusted for visual acuity at randomization; Test type: Superiority; Mean Difference (Final Values) = -2, 98.3% CI 2-sided [-13 to 9]

10. Secondary Outcome: VA Improvement at 8 Weeks Defined as a Binary Outcome
Description: A secondary analysis will estimate the proportion of subjects with amblyopic-eye VA improvement of ≥ 2 logMAR lines (≥ 10 letters if E-ETDRS) at 8 weeks after baseline.
Time Frame: At 8 weeks
Population: Of 68 participants in the continued spectacle correction older cohort, only 67 visits were completed in the analysis window.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 67 | 85 | 84
Participants | 5 | 6 | 35 | 25
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Binomial regression was used for the treatment group comparison of the proportion of participants classified as improving 2 or more logMAR lines (10 or more letters if E-ETDRS) from baseline at the 8-week visit, adjusted for visual acuity at randomization; Test type: Superiority; Mean Difference (Final Values) = -1, 98.3% CI 2-sided [-15 to 12]; For secondary visual acuity outcomes, which included the 8-week treatment group comparison, a Bonferroni adjustment was used to control for multiple testing (3 outcomes tested) to preserve the overall type I error rate at 5% (2-sided alpha=0.017 per test)

11. Secondary Outcome: Distribution of Stereoacuity Scores at 4 Weeks
Description: Stereoacuity will be tested at near in current refractive correction using the Randot Butterfly and Randot Preschool stereoacuity tests. Stereoacuity scores (measure as seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods.
  Lower scores indicate better stereoacuity. Results of the Randot Butterfly test were analyzed as 2000 seconds of arc (if correct response). Nil was assigned a score of 4000 seconds of arc and was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted.
Time Frame: 4 weeks
Population: Limited to those with follow-up visits completed within the pre-specified analysis window
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 85 | 84
Participants
  Missing/Not done | 0 | 0 | 6 | 8
  Nil | 31 | 25 | 24 | 21
  2000 | 11 | 11 | 8 | 10
  800 | 9 | 5 | 13 | 7
  400 | 7 | 6 | 10 | 15
  200 | 3 | 5 | 9 | 9
  100 | 4 | 12 | 10 | 6
  60 | 2 | 2 | 3 | 5
  40 | 2 | 1 | 2 | 3

12. Secondary Outcome: Distribution of Change in Stereoacuity Scores From Baseline
Description: Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods. Lower scores indicate better stereoacuity. Results of the Randot Butterfly test were analyzed as 2000 (if correct response). Nil (4000) was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted. For each visit, stereoacuity scores were ordered and assigned a rank score. Change in stereoacuity was calculated as the difference in ranked score between the enrollment and 4-week stereoacuity scores.
Time Frame: 4 weeks
Population: Change was only calculated if data was available at both baseline and 4 week time points. Some baseline data was missing in the younger cohort, leading to the numerical inconsistency.
Measure: Count of Participants; unit: Participants
Groups:
- Continued Spectacle Correction Younger Cohort: Binocular computer game treatment is defined as playing a Dig Rush application on an iPad® 1 hour per day, 5 days per week for 8 weeks in addition to continued spectacle correction (if required)
  iPad®: Binocular therapy using a Dig Rush application on an iPad®
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 78 | 73
Participants
  2 or more levels worse | 8 | 6 | 11 | 8
  Within 1 level | 53 | 50 | 56 | 57
  2 or more levels better | 8 | 11 | 11 | 8
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Test type: Superiority; p = 0.38, Wilcoxon (Mann-Whitney) — The exact Wilcoxon rank-sum test was used to compare the change in stereoacuity levels from baseline to the 4-week visit by treatment group

13. Secondary Outcome: Distribution of Stereoacuity Scores at 8 Weeks
Description: as for outcome 11
Time Frame: 8 weeks
Population: Limited to those with follow-up visits completed within the pre-specified analysis window
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 85 | 84
Participants
  Nil | 31 | 24 | 28 | 25
  2000 | 11 | 10 | 11 | 8
  800 | 5 | 8 | 10 | 15
  400 | 4 | 2 | 9 | 12
  200 | 5 | 11 | 12 | 9
  100 | 6 | 9 | 10 | 7
  60 | 2 | 3 | 2 | 3
  40 | 3 | 1 | 3 | 5

14. Secondary Outcome: Distribution of Change in Stereoacuity Scores From Baseline
Description: Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods. Lower scores indicate better stereoacuity. Results of the Randot Butterfly test were analyzed as 2000 (if correct response). Nil (4000) was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted. For each visit, stereoacuity scores were ordered and assigned a rank score. Change in stereoacuity was calculated as the difference in ranked score between the enrollment and 8-week stereoacuity scores.
Time Frame: 8 weeks
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 85 | 72
Participants
  2 or more levels worse | 6 | 3 | 8 | 3
  Within 1 level | 53 | 51 | 65 | 54
  2 or more levels better | 8 | 14 | 12 | 15
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney) — The exact Wilcoxon rank-sum test was used to compare the change in stereoacuity levels from baseline to the 8-week visit by treatment group

15. Secondary Outcome: Distribution of Stereoacuity Scores (Participants With no History of Strabismus)
Description: Stereoacuity was tested at near in current refractive correction. Stereoacuity scores (measure as seconds of arc) were calculated based on the Randot Butterfly (scores: 2000, Nil) and Randot Preschool stereoacuity (scores: 800, 400, 200, 100, 60 and 40) test methods.
  Lower scores indicate better stereoacuity. Results of the Randot Butterfly test were analyzed as 2000 seconds of arc (if correct response). Nil was assigned a score of 4000 seconds of arc and was defined as (1) an incorrect response on the butterfly in absence of a correct response on the 800 seconds of arc level of the Randot Preschool stereoacuity test or (2) an incorrect response on the 800 seconds of arc level if the butterfly was not attempted.
Time Frame: 4 weeks
Population: Only participants with no history of strabismus are analyzed, as mentioned in the outcome title.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 27 | 37 | 58 | 51
Participants
  Missing/Not Done | 0 | 0 | 4 | 4
  Nil | 8 | 7 | 11 | 8
  2000 | 3 | 5 | 5 | 7
  800 | 2 | 3 | 8 | 4
  400 | 5 | 4 | 8 | 10
  200 | 1 | 4 | 9 | 9
  100 | 4 | 12 | 10 | 4
  60 | 2 | 1 | 3 | 4
  40 | 2 | 1 | 0 | 1

16. Secondary Outcome: Distribution of Change in Stereoacuity Scores From Baseline (Participants With no History of Strabismus)
Description: as for outcome 12
Time Frame: 4 weeks
Population: Only participants with no history of strabismus are analyzed, as mentioned in the outcome title. Change was only calculated if data was available at both baseline and 4 week time points. Some baseline data was missing in the younger cohort, leading to the numerical inconsistency.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 27 | 37 | 54 | 45
Participants
  2 or more levels worse | 5 | 2 | 8 | 6
  Within 1 level | 17 | 27 | 37 | 34
  2 or more levels better | 5 | 8 | 9 | 5
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Test type: Superiority; p = 0.19, Wilcoxon (Mann-Whitney) — The exact Wilcoxon rank-sum test was used to compare the change in stereoacuity levels from baseline to the 4-week visit by treatment group for participants without strabismus

17. Secondary Outcome: Distribution of Stereoacuity Scores (Participants With no History of Strabismus)
Description: as for outcome 15
Time Frame: 8 weeks
Population: Only participants with no history of strabismus are analyzed, as mentioned in the outcome title.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 27 | 38 | 57 | 51
Participants
  Nil | 8 | 8 | 14 | 11
  2000 | 3 | 7 | 8 | 4
  800 | 1 | 1 | 5 | 8
  400 | 1 | 1 | 5 | 8
  200 | 5 | 9 | 11 | 8
  100 | 4 | 9 | 9 | 6
  60 | 2 | 3 | 2 | 2
  40 | 3 | 0 | 3 | 4

18. Secondary Outcome: Distribution of Change in Stereoacuity Scores From Baseline (Participants With no History of Strabismus)
Description: as for outcome 12
Time Frame: 8 weeks
Population: Only participants with no history of strabismus are analyzed, as mentioned in the outcome title.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 27 | 38 | 57 | 51
Participants
  2 or more levels worse | 3 | 0 | 5 | 4
  Within 1 level | 19 | 31 | 44 | 34
  2 or more levels better | 5 | 7 | 8 | 13
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney) — The exact Wilcoxon rank-sum test was used to compare the change in stereoacuity levels from baseline to the 8-week visit by treatment group for participants without strabismus

19. Secondary Outcome: Binocular Therapy: Treatment Compliance and Fellow-Eye Contrast
Description: Data from the automated iPad log files will be used to provide an objective measure of compliance with binocular treatment (participants completion of >75% of prescribed game play). The total amount of game play will be computed for the initial 4 weeks of treatment for the binocular treatment group, as well as throughout 8 weeks. Secondary analyses will evaluate the relationship between the total amount of game play with (1) change in VA and (2) change in stereoacuity after the first 4 weeks of binocular treatment. Data from the automated iPad log files will also be used to assess game performance as measured by the fellow-eye contrast.
Time Frame: 4 weeks
Population: The control group was not prescribed binocular therapy, which is why they were not included here.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Binocular Computer Game Treatment Younger Cohort
Number analyzed (Participants) | 69 | 84
Participants
  Completed >75% prescribed game play | 40 | 37
  Fellow-eye contrast of 100% | 30 | 32
  Fellow-eye contrast of 20% or worse | 1 | 3

20. Secondary Outcome: Binocular Therapy: Treatment Compliance and Fellow-Eye Contrast
Description: Data from the automated iPad log files will be used to assess game performance as measured by the fellow-eye contrast. The level and change in fellow-eye contrast will be computed for the initial 4 weeks of treatment for the binocular treatment group. Secondary analyses will evaluate the relationship between the change in fellow-eye contrast with (1) change in VA and (2) change in stereoacuity after the first 8 weeks of binocular treatment. Data from the automated iPad log files will also be used to assess game performance as measured by the fellow-eye contrast.
Time Frame: 8 weeks
Population: Data from automated iPad log files were only able to be retrieved successfully for 81 of 85 participants in the younger cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Binocular Computer Game Treatment Younger Cohort
Number analyzed (Participants) | 67 | 81
Participants
  Completed >75% prescribed game play | 38 | 35
  Fellow-eye contrast of 100% | 59 | 50
  Fellow-eye contrast of 20% or worse | 1 | 2

21. Secondary Outcome: Treatment Compliance With Spectacle Wear
Description: Parent-reported adherence with spectacle wear (excluding participants with reported compliance of 'N/A') for the initial 4 weeks. Patient reported to have completed >75% of spectacle wear at 4 weeks.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 85 | 78
Participants | 57 | 57 | 66 | 74

22. Secondary Outcome: Treatment Compliance With Spectacle Wear
Description: Parent-reported adherence with spectacle wear (excluding participants with reported compliance of 'N/A') across 8 weeks. Patient reported to have completed >75% of spectacle wear at 8 weeks.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 89 | 82
Participants | 61 | 62 | 69 | 78

23. Secondary Outcome: Mean Change in Fellow Eye Visual Acuity at 4 Weeks (Older Cohort)
Description: The mean change in fellow-eye VA from baseline to 4 weeks will be calculated and compared between treatment groups using ANCOVA with adjustment for baseline VA.
Time Frame: Baseline and 4 weeks
Measure: Mean (99% Confidence Interval); unit: Letters
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort
Number analyzed (Participants) | 69 | 67
Letters
  Adjusted | 0.1 [-1.1 to 1.1] | 1.1 [0.1 to 2.2]
  Unadjusted | 0.1 [-1.1 to 1.3] | 1.1 [0.2 to 2.1]
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; An analysis of covariance (ANCOVA) model was used to compute the treatment group difference in the mean change in fellow-eye visual acuity (letters) from baseline to 4 weeks, adjusting for fellow-eye visual acuity at randomization. A 2-sided 99% confidence interval was computed on the adjusted treatment group difference; Test type: Superiority; Mean Difference (Final Values) = -1.1, 99% CI 2-sided [-2.5 to 0.4] — Statistical significance of the treatment group comparison was based on a 2-sided alpha=0.01

24. Secondary Outcome: Mean Change in Fellow Eye VA at 8 Weeks (Older Cohort)
Description: The mean change in fellow-eye VA from baseline to 8 weeks will be calculated and compared between treatment groups using ANCOVA with adjustment for baseline VA.
Time Frame: Baseline and 8 weeks
Measure: Mean (99% Confidence Interval); unit: Letters
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort
Number analyzed (Participants) | 68 | 67
Letters
  Adjusted | 0.5 [-0.5 to 1.4] | 1.5 [0.5 to 2.4]
  Unadjusted | 0.5 [-0.6 to 1.6] | 1.5 [0.7 to 2.3]
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; An analysis of covariance (ANCOVA) model was used to compute the treatment group difference in the mean change in fellow-eye visual acuity (letters) from baseline to 8 weeks, adjusting for fellow-eye visual acuity at randomization. A 2-sided 99% confidence interval was computed on the adjusted treatment group difference; Test type: Superiority; Mean Difference (Final Values) = -1.0, 99% CI 2-sided [-2.3 to 0.3] — Statistical significance of the treatment group comparison was based on a 2-sided alpha=0.01

25. Secondary Outcome: Ocular Alignment at 4 Weeks
Description: The proportion of subjects with development of new strabismus (no heterotropia at baseline and the presence of near and/or distance heterotropia at 4 weeks) or an increase from baseline ≥10∆ in a pre-existing strabismus at 4 weeks will be reported by treatment group and compared using Barnard's exact test.
  Ocular alignment will be assessed in current refractive correction by the cover/uncover test, simultaneous prism and cover test (SPCT), and prism and alternate cover test (PACT) in primary gaze at distance (3 meters) and at near (1/3 meter).
  Participants were classified according to whether they met the any of the following criteria at the 4-week visit: development of a new tropia (measured by SPCT) and/or worsening of a pre-existing deviation by 10 prism diopters (pd) measured by SPCT.
Time Frame: 4 weeks
Population: As this was a safety outcome, all visit information was recorded, regardless of whether or not it was collected in the analysis window.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 88 | 84
Participants | 10 | 6 | 7 | 7
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Fisher's exact test was used to perform the treatment group comparison of the proportion of participants who developed a new ocular deviation and/or worsening of a pre-existing ocular deviation by 10 prism diopters at the 4-week visit; Test type: Superiority; p = 0.37, Fisher Exact

26. Secondary Outcome: Ocular Alignment at 8 Weeks
Description: The proportion of subjects with development of new strabismus (no heterotropia at baseline and the presence of near and/or distance heterotropia at 8 weeks) or an increase from baseline ≥10∆ in a pre-existing strabismus at 8 weeks will be reported by treatment group and compared using Barnard's exact test.
  Ocular alignment will be assessed in current refractive correction by the cover/uncover test, simultaneous prism and cover test (SPCT), and prism and alternate cover test (PACT) in primary gaze at distance (3 meters) and at near (1/3 meter).
  Participants were classified according to whether they met the any of the following criteria at the 8-week visit: development of a new tropia (measured by SPCT) and/or worsening of a pre-existing deviation by 10 prism diopters (pd) measured by SPCT.
Time Frame: 8 weeks
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 86 | 84
Participants | 9 | 9 | 6 | 7
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; Fisher's exact test was used to perform the treatment group comparison of the proportion of participants who developed a new ocular deviation and/or worsening of a pre-existing ocular deviation by 10 prism diopters at the 8-week visit; Test type: Superiority; p = 0.99, Fisher Exact

27. Secondary Outcome: Distribution of Diplopia Frequency at 4 Weeks (Participant-reported)
Description: The proportion of subjects with each level of diplopia frequency will be reported by treatment group at 4 weeks.
  A standardized questionnaire was administered to participants and their parents to assess the presence and frequency of any diplopia since the last study visit.
Time Frame: 4 weeks
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 87 | 84
Participants
  Never | 62 | 64 | 78 | 79
  Less than once a week | 1 | 0 | 2 | 2
  Once a week | 2 | 2 | 4 | 0
  Once a day | 2 | 1 | 3 | 3
  Up to 10 times a day | 2 | 0 | 0 | 0
  More than 10 times a day | 0 | 0 | 0 | 0
  All the time | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; The frequency of diplopia, across categories of diplopia, was compared between the treatment groups using the Cochran-Armitage trend test; Test type: Superiority; p = 0.20, Cochran-Armitage trend test

28. Secondary Outcome: Distribution of Diplopia Frequency at 8 Weeks (Participant-reported)
Description: The proportion of subjects with each level of diplopia frequency will be reported by treatment group at 8 weeks.
  A standardized questionnaire was administered to participants and their parents to assess the presence and frequency of any diplopia since the last study visit.
Time Frame: 8 weeks
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 68 | 68 | 86 | 84
Participants
  Never | 63 | 65 | 78 | 78
  Less than once a week | 5 | 2 | 4 | 4
  Once a week | 0 | 0 | 1 | 1
  Once a day | 0 | 1 | 2 | 0
  Up to 10 times a day | 0 | 0 | 1 | 0
  More than 10 times a day | 0 | 0 | 0 | 0
  All the time | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p > 0.99, Cochran-Armitage trend test

29. Secondary Outcome: Change in Diplopia Frequency From Baseline to 4 Weeks (Participant-reported)
Description: A standardized questionnaire was administered to participants and their parents to assess the presence and frequency of any diplopia since the last study visit. Change in diplopia frequency from baseline to 4 weeks was reported categorically.
Time Frame: 4 weeks
Population: As this was a safety outcome, all visit information was recorded, regardless of whether or not it was collected in the analysis window. There was 1 missing participant-reported diplopia frequency at baseline in the Binocular Younger cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 86 | 84
Participants
  Increased frequency (≥ 2 levels) | 3 | 2 | 6 | 2
  Similar frequency (within 1 level) | 64 | 64 | 79 | 80
  Reduced frequency (≥ 2 levels) | 2 | 1 | 1 | 2
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; The exact Wilcoxon rank-sum test was used to compare the change in diplopia frequency levels from baseline to the 4-week visit by treatment group; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Change in Diplopia Frequency From Baseline to 8 Weeks (Participant-reported)
Description: A standardized questionnaire was administered to participants and their parents to assess the presence and frequency of any diplopia since the last study visit. Change in diplopia frequency from baseline to 8 weeks was reported categorically.
Time Frame: 8 weeks
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 68 | 68 | 85 | 84
Participants
  Increased frequency (≥ 2 levels) | 0 | 1 | 2 | 1
  Similar frequency (within 1 level) | 64 | 66 | 82 | 80
  Reduced frequency (≥ 2 levels) | 4 | 1 | 1 | 3
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; The exact Wilcoxon rank-sum test was used to compare the change in diplopia frequency levels from baseline to the 8-week visit by treatment group; Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: Distribution of Diplopia Frequency at 4 Weeks (Parent-reported)
Description: as for outcome 27
Time Frame: 4 weeks
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 66 | 88 | 83
Participants
  Never | 65 | 66 | 87 | 83
  Less than once a week | 3 | 0 | 1 | 0
  Once a week | 1 | 0 | 0 | 0
  Once a day | 0 | 0 | 0 | 0
  Up to 10 times a day | 0 | 0 | 0 | 0
  More than 10 times a day | 0 | 0 | 0 | 0
  All the time | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p = 0.12, Cochran-Armitage trend test

32. Secondary Outcome: Distribution of Diplopia Frequency at 8 Weeks (Parent-reported)
Description: as for outcome 28
Time Frame: 8 weeks
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 86 | 84
Participants
  Never | 66 | 67 | 84 | 84
  Less than once a week | 1 | 1 | 2 | 0
  Once a week | 0 | 0 | 0 | 0
  Once a day | 0 | 0 | 0 | 0
  Up to 10 times a day | 0 | 0 | 0 | 0
  More than 10 times a day | 0 | 0 | 0 | 0
  All the time | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p > 0.99, Cochran-Armitage trend test

33. Secondary Outcome: Change in Diplopia Frequency From Baseline to 4 Weeks (Parent-reported)
Description: as for outcome 29
Time Frame: 4 weeks
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 66 | 88 | 83
Participants
  Increased frequency (≥ 2 levels) | 0 | 0 | 0 | 0
  Similar frequency (within 1 level) | 69 | 66 | 88 | 82
  Reduced frequency (≥ 2 levels) | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

34. Secondary Outcome: Change in Diplopia Frequency From Baseline to 8 Weeks (Parent-reported)
Description: as for outcome 30
Time Frame: 8 weeks
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 86 | 84
Participants
  Increased frequency (≥ 2 levels) | 0 | 0 | 0 | 0
  Similar frequency (within 1 level) | 67 | 68 | 86 | 83
  Reduced frequency (≥ 2 levels) | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; [analysis description as in outcome 30, analysis 1]; Test type: Superiority; p > 0.99, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Frequency of Adverse Symptoms (Symptom Survey)
Description: The child and parent(s) will complete a 5-item symptom survey regarding the presence of various ocular symptoms within the past 2 weeks at enrollment and at each visit. The distribution of scores on each symptom survey item will be described for the enrollment exam and the 4-week exam for each treatment group. The distribution of change in scores on each symptom survey item will also be described for each treatment group.
Time Frame: 4 weeks
Population: There were 3 participants in the older cohort control treatment group with responses of 'Not wearing spectacles'. These participants were excluded from the percentage tabulations (only the number is reported) in the table and any analyses specific to these Symptom Survey items.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 88 | 83
Participants
  Blurred Vision: Never | 61 | 57 | 72 | 71
  Blurred Vision: Almost Never | 3 | 8 | 10 | 6
  Blurred Vision: Sometimes | 5 | 1 | 5 | 4
  Blurred Vision: Often | 0 | 1 | 1 | 2
  Blurred Vision: Almost Always | 0 | 0 | 0 | 0
  Eyestrain: Never | 50 | 46 | 53 | 58
  Eyestrain: Almost Never | 7 | 13 | 15 | 19
  Eyestrain: Sometimes | 9 | 7 | 17 | 6
  Eyestrain: Often | 2 | 1 | 3 | 0
  Eyestrain: Almost Always | 1 | 0 | 0 | 0
  Headache: Never | 38 | 38 | 60 | 68
  Headache: Almost Never | 20 | 14 | 14 | 13
  Headache: Sometimes | 8 | 12 | 9 | 1
  Headache: Often | 3 | 3 | 5 | 1
  Headache: Almost Always | 0 | 0 | 0 | 0
  Look Over Spectacles: number analyzed (Participants) | 69 | 64 | 88 | 83
  Look Over Spectacles: Never | 44 | 39 | 44 | 40
  Look Over Spectacles: Almost Never | 11 | 9 | 17 | 19
  Look Over Spectacles: Sometimes | 13 | 11 | 19 | 17
  Look Over Spectacles: Often | 1 | 5 | 6 | 6
  Look Over Spectacles: Almost Always | 0 | 0 | 2 | 1
  Take Off Spectacles: number analyzed (Participants) | 69 | 64 | 88 | 83
  Take Off Spectacles: Never | 43 | 41 | 43 | 46
  Take Off Spectacles: Almost Never | 13 | 14 | 26 | 24
  Take Off Spectacles: Sometimes | 12 | 9 | 15 | 11
  Take Off Spectacles: Often | 1 | 0 | 4 | 1
  Take Off Spectacles: Almost Always | 0 | 0 | 0 | 1

36. Secondary Outcome: Frequency of Adverse Symptoms (Symptom Survey) at 8 Weeks
Description: as for outcome 35
Time Frame: 8 weeks
Population: There were 3 participants in the control treatment group with responses of 'Not wearing spectacles'. These participants were excluded from the percentage tabulations (only the number is reported) in the table and any analyses specific to these Symptom Survey items.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 86 | 84
Participants
  Blurred Vision: Never | 58 | 61 | 74 | 62
  Blurred Vision: Almost Never | 7 | 4 | 5 | 17
  Blurred Vision: Sometimes | 2 | 2 | 7 | 5
  Blurred Vision: Often | 0 | 1 | 0 | 0
  Blurred Vision: Almost Always | 0 | 0 | 0 | 0
  Eyestrain: Never | 48 | 47 | 58 | 58
  Eyestrain: Almost Never | 9 | 13 | 16 | 20
  Eyestrain: Sometimes | 9 | 7 | 12 | 6
  Eyestrain: Often | 1 | 1 | 0 | 0
  Eyestrain: Almost Always | 0 | 0 | 0 | 0
  Headache: Never | 44 | 44 | 62 | 65
  Headache: Almost Never | 13 | 17 | 13 | 17
  Headache: Sometimes | 8 | 6 | 10 | 2
  Headache: Often | 2 | 1 | 1 | 0
  Headache: Almost Always | 0 | 0 | 0 | 0
  Look Over Spectacles: number analyzed (Participants) | 67 | 65 | 86 | 84
  Look Over Spectacles: Never | 42 | 41 | 38 | 40
  Look Over Spectacles: Almost Never | 15 | 11 | 16 | 17
  Look Over Spectacles: Sometimes | 9 | 10 | 26 | 23
  Look Over Spectacles: Often | 1 | 2 | 5 | 2
  Look Over Spectacles: Almost Always | 0 | 1 | 1 | 2
  Take Off Spectacles: number analyzed (Participants) | 67 | 65 | 86 | 84
  Take Off Spectacles: Never | 40 | 43 | 45 | 44
  Take Off Spectacles: Almost Never | 16 | 17 | 28 | 30
  Take Off Spectacles: Sometimes | 10 | 4 | 8 | 7
  Take Off Spectacles: Often | 0 | 1 | 5 | 3
  Take Off Spectacles: Almost Always | 1 | 0 | 0 | 0

37. Secondary Outcome: Distribution of Change in Adverse Symptom Frequency (Symptom Survey) From Baseline to 4 Weeks
Description: as for outcome 35
Time Frame: 4 weeks
Population: There were 3 participants in the control treatment group with responses of 'Not wearing spectacles'. These participants were excluded from the tabulations in the table and any analyses specific to these Symptom Survey items.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 88 | 83
Participants
  Blurred Vision: Increased frequency (≥ 2 levels) | 1 | 1 | 4 | 0
  Blurred Vision: Similar frequency (within 1 level) | 62 | 59 | 73 | 72
  Blurred Vision: Reduced frequency (≥ 2 levels) | 6 | 7 | 11 | 11
  Eyestrain: Increased frequency (≥ 2 levels) | 1 | 3 | 9 | 0
  Eyestrain: Similar frequency (within 1 level) | 61 | 52 | 73 | 73
  Eyestrain: Reduced frequency (≥ 2 levels) | 7 | 12 | 6 | 10
  Headache: Increased frequency (≥ 2 levels) | 2 | 2 | 7 | 0
  Headache: Similar frequency (within 1 level) | 60 | 58 | 76 | 72
  Headache: Reduced frequency (≥ 2 levels) | 7 | 7 | 5 | 11
  Look Over Spectacles: number analyzed (Participants) | 69 | 64 | 88 | 83
  Look Over Spectacles: Increased frequency (≥ 2 levels) | 2 | 5 | 4 | 2
  Look Over Spectacles: Similar frequency (within 1 level) | 60 | 46 | 72 | 73
  Look Over Spectacles: Reduced frequency (≥ 2 levels) | 7 | 13 | 12 | 8
  Take Off Spectacles: number analyzed (Participants) | 69 | 64 | 88 | 83
  Take Off Spectacles: Increased frequency (≥ 2 levels) | 0 | 0 | 1 | 0
  Take Off Spectacles: Similar frequency (within 1 level) | 64 | 54 | 78 | 80
  Take Off Spectacles: Reduced frequency (≥ 2 levels) | 5 | 10 | 9 | 3
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort vs Binocular Computer Game Treatment Younger Cohort vs Continued Spectacle Correction Younger Cohort; For each Symptom Survey item, the exact Wilcoxon rank-sum test was used to compare the change in symptom frequency level from baseline to the 4-week visit by treatment group; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)

38. Secondary Outcome: Distribution of Change in Adverse Symptom Frequency (Symptom Survey) From Baseline to 8 Weeks
Description: The child and parent(s) will complete a 5-item symptom survey regarding the presence of various ocular symptoms within the past 2 weeks at enrollment and at each visit. The distribution of scores on each symptom survey item will be described for the enrollment exam and the 8-week exam for each treatment group. The distribution of change in scores on each symptom survey item will also be described for each treatment group.
Time Frame: 8 weeks
Population: There were 3 participants in the control treatment group with responses of 'Not wearing spectacles'. These participants were excluded from the tabulations in the table and any analyses specific to these Symptom Survey items. One participant in the binocular treatment group did not have a completed Symptom Survey at the 8-week visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 67 | 68 | 86 | 84
Participants
  Blurred Vision: Increased frequency (≥ 2 levels) | 1 | 2 | 4 | 2
  Blurred Vision: Similar frequency (within 1 level) | 61 | 57 | 67 | 71
  Blurred Vision: Reduced frequency (≥ 2 levels) | 5 | 9 | 15 | 11
  Eyestrain: Increased frequency (≥ 2 levels) | 1 | 1 | 5 | 1
  Eyestrain: Similar frequency (within 1 level) | 60 | 55 | 75 | 72
  Eyestrain: Reduced frequency (≥ 2 levels) | 6 | 12 | 6 | 11
  Headache: Increased frequency (≥ 2 levels) | 2 | 0 | 5 | 0
  Headache: Similar frequency (within 1 level) | 60 | 59 | 76 | 77
  Headache: Reduced frequency (≥ 2 levels) | 5 | 9 | 5 | 7
  Look Over Spectacles: number analyzed (Participants) | 67 | 65 | 86 | 84
  Look Over Spectacles: Increased frequency (≥ 2 levels) | 3 | 0 | 6 | 3
  Look Over Spectacles: Similar frequency (within 1 level) | 54 | 50 | 70 | 76
  Look Over Spectacles: Reduced frequency (≥ 2 levels) | 10 | 15 | 10 | 5
  Take Off Spectacles: number analyzed (Participants) | 67 | 65 | 86 | 84
  Take Off Spectacles: Increased frequency (≥ 2 levels) | 0 | 0 | 0 | 2
  Take Off Spectacles: Similar frequency (within 1 level) | 62 | 55 | 76 | 77
  Take Off Spectacles: Reduced frequency (≥ 2 levels) | 5 | 10 | 10 | 5
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort vs Binocular Computer Game Treatment Younger Cohort vs Continued Spectacle Correction Younger Cohort; For each Symptom Survey item, the exact Wilcoxon rank-sum test was used to compare the change in symptom frequency level from baseline to the 8-week visit by treatment group. This was utilized for each item in the survey; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)

39. Secondary Outcome: Mean Change in Fellow Eye Visual Acuity at 4 Weeks (Younger Cohort)
Description: as for outcome 23
Time Frame: Baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: logMAR Lines
Arm/Group | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 88 | 84
logMAR Lines
  Adjusted | 0.0536 [-0.1 to 0.2] | 0.1939 [0.02 to 0.4]
  Unadjusted | 0.0682 [-0.1 to 0.2] | 0.1786 [0.02 to 0.4]

40. Secondary Outcome: Mean Change in Fellow Eye VA at 8 Weeks (Younger Cohort)
Description: as for outcome 24
Time Frame: baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: logMAR Lines
Arm/Group | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 86 | 84
logMAR Lines
  Adjusted | 0.3160 [0.1 to 0.5] | 0.2122 [0.04 to 0.4]
  Unadjusted | 0.3256 [0.1 to 0.5] | 0.2024 [-0.1 to 0.3]

41. Other Pre Specified Outcome: Exploratory Analysis: Subgroup VA Change Analysis at 4 Weeks
Description: The treatment effect after 4 weeks in subgroups based on baseline factors will be assessed in exploratory analyses and used to suggest hypotheses for further investigation in future studies. The following baseline factors are of interest: amblyopic-eye VA, stereoacuity, the presence of a tropia at near, and prior amblyopia treatment (other than spectacle correction). In accordance with NIH guidelines, subgroup analyses of treatment effect according to gender and race/ethnicity will be conducted. Positive values for visual acuity change indicate improvement.
Time Frame: Baseline and 4 weeks
Population: Analyses were limited to participants who completed the 4-week visit within the pre-defined analysis window (21 to <49 days after randomization).
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
Number analyzed (Participants) | 69 | 67 | 85 | 84
Letters
  Overall | 1.3 (5.3) | 1.7 (5.5) | 1.1 (1.4) | 0.6 (1.3)
  Sex: Female: number analyzed (Participants) | 30 | 34 | 47 | 43
  Sex: Female | 1.5 (4.6) | 1.8 (6.0) | 1.2 (1.4) | 0.7 (1.4)
  Sex: Male: number analyzed (Participants) | 39 | 33 | 38 | 41
  Sex: Male | 1.2 (5.8) | 1.6 (4.9) | 1.0 (1.4) | 0.5 (1.1)
  Age at Randomization: 4 to <5: number analyzed (Participants) | 0 | 0 | 10 | 16
  Age at Randomization: 4 to <5 |  |  | 0.8 (1.2) | 0.8 (1.2)
  Age at Randomization: 5 to <7: number analyzed (Participants) | 0 | 0 | 75 | 68
  Age at Randomization: 5 to <7 |  |  | 1.1 (1.5) | 0.6 (1.3)
  Age at Randomization: 7 to <10: number analyzed (Participants) | 45 | 43 | 0 | 0
  Age at Randomization: 7 to <10 | 1.6 (6.0) | 2.0 (5.4) |  |
  Age at Randomization: 10 to <13: number analyzed (Participants) | 24 | 24 | 0 | 0
  Age at Randomization: 10 to <13 | 0.9 (3.8) | 1.2 (5.6) |  |
  Race: Non-white/Hispanic: number analyzed (Participants) | 19 | 14 | 16 | 13
  Race: Non-white/Hispanic | 2.5 (6.8) | 3.7 (7.2) | 1.1 (1.3) | 0.5 (0.8)
  Race: White/Non-Hispanic: number analyzed (Participants) | 50 | 53 | 69 | 71
  Race: White/Non-Hispanic | 0.9 (4.6) | 1.2 (4.8) | 1.1 (1.5) | 0.6 (1.3)
  Baseline VA: 20/080 to 20/200: number analyzed (Participants) | 23 | 29 | 21 | 18
  Baseline VA: 20/080 to 20/200 | 3.2 (5.9) | 1.3 (6.5) | 1.0 (1.3) | 0.7 (1.4)
  Baseline VA: 20/063: number analyzed (Participants) | 19 | 13 | 22 | 23
  Baseline VA: 20/063 | 1.5 (3.7) | 2.5 (5.5) | 0.9 (1.5) | 0.5 (1.2)
  Baseline VA: 20/050: number analyzed (Participants) | 11 | 10 | 25 | 25
  Baseline VA: 20/050 | 1.6 (4.2) | 0.9 (3.3) | 1.4 (1.5) | 0.5 (1.1)
  Baseline VA: 20/040: number analyzed (Participants) | 16 | 15 | 17 | 18
  Baseline VA: 20/040 | -1.7 (5.9) | 2.2 (4.5) | 1.1 (1.5) | 0.9 (1.4)
  Prior Amblyopia Treatment: No: number analyzed (Participants) | 4 | 2 | 32 | 28
  Prior Amblyopia Treatment: No | 0.5 (3.0) | 5.0 (5.7) | 0.9 (1.1) | 0.6 (1.1)
  Prior Amblyopia Treatment: Yes: number analyzed (Participants) | 65 | 65 | 53 | 56
  Prior Amblyopia Treatment: Yes | 1.4 (5.4) | 1.6 (5.5) | 1.2 (1.6) | 0.6 (1.4)
  Prior Binocular Treatment: No: number analyzed (Participants) | 68 | 64 | 0 | 0
  Prior Binocular Treatment: No | 1.3 (5.3) | 2.2 (5.2) |  |
  Prior Binocular Treatment: Yes: number analyzed (Participants) | 1 | 3 | 0 | 0
  Prior Binocular Treatment: Yes | 3.0 (0) | -5.8 (3.1) |  |
  Baseline stereoacuity at near: Nil: number analyzed (Participants) | 33 | 31 | 27 | 26
  Baseline stereoacuity at near: Nil | 1.6 (5.5) | 0.7 (5.6) | 0.9 (1.6) | 0.3 (1.2)
  Baseline stereoacuity at near: Better than Nil: number analyzed (Participants) | 36 | 36 | 58 | 57
  Baseline stereoacuity at near: Better than Nil | 1.1 (5.2) | 2.5 (5.2) | 1.2 (1.4) | 0.8 (1.3)
  Near Heterotropia at Randomization: No: number analyzed (Participants) | 44 | 45 | 66 | 70
  Near Heterotropia at Randomization: No | 2.0 (5.2) | 2.2 (5.6) | 1.1 (1.5) | 0.7 (1.3)
  Near Heterotropia at Randomization: Yes: number analyzed (Participants) | 25 | 22 | 19 | 14
  Near Heterotropia at Randomization: Yes | 0.1 (5.4) | 0.7 (5.1) | 1.1 (1.2) | 0.4 (1.3)
Statistical Analysis 1: Comparison: Binocular Computer Game Treatment Older Cohort vs Continued Spectacle Correction Older Cohort; An analysis of covariance (ANCOVA) was performed to test the 2-way interaction between treatment group with each factor (baseline age and visual acuity were treated as continuous factors), adjusting for baseline amblyopic-eye visual acuity and the nested terms from the interaction term. Formal subgroup analyses were only performed if there was a minimum of 20 participants in every subgroup category across both treatment groups for factors treated as categorical variables in the model; Test type: Superiority; p > 0.01, ANCOVA — Statistical significance of the interaction term was based on a 2-sided alpha=0.01

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Binocular Computer Game Treatment Older Cohort | Continued Spectacle Correction Older Cohort | Binocular Computer Game Treatment Younger Cohort | Continued Spectacle Correction Younger Cohort
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69 | 0/92 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69 | 0/92 | 0/90
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69 | 0/92 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02983552/Prot_001.pdf
  • Statistical Analysis Plan (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02983552/SAP_002.pdf
  • Informed Consent Form (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02983552/ICF_000.pdf